CLINICAL TRIAL: NCT01674296
Title: Seasonality of Stress, Diet, and Physical Activity in Mid-Life Women
Brief Title: Seasonal Patterns of Stress, Diet and Physical Activity - Life in All Seasons (LENAS)
Acronym: LENAS
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC018
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Stress; Feeding Behavior; Physical Activity
Keywords: Body Weight/physiology*; Diet*/statistics & numerical data; Diet*/trends; Exercise/physiology*; Female; Humans; Longitudinal Studies; Middle Aged; Obesity/epidemiology*; Seasons*; Time Factors
MeSH Terms: conditions — Obesity; Feeding Behavior; Motor Activity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Buffy Coat, Urine, Saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 (2012-2013): Monitoring of Dietary Intake, Physical Activity and Stress
- Group 2 (2013-2014): Monitoring of Dietary Intake, Physical Activity and Stress

SUMMARY:
The purpose of this study is to develop a better understanding of factors affecting American's energy balance related behaviors - in this case, food intake and activity. In the present study we will describe the relative contributions of individual psychology and physiology (including metabolism, mood, and sleep habits) and external (season, stressors) contributions to changes in adiposity over a year in free-living individuals.

This study will illuminate season's role in changes in energy balance related behaviors and body weight and composition. Ultimately, this information will be used to identify factors affecting food consumption and individual activity during seasonal periods to help to segment interventions for obesity prevention in mid-life women.

DETAILED DESCRIPTION:
This is a longitudinal, observational study of mid-life women spanning one year.There will be frequent monitoring of food consumption, individual activity and individual- level factors thought to influence food consumption and activity such as dietary restraint, subjective stress, sleep quality and duration, and physiological stress as measured by allostatic load.

Specific aims:

1. To identify seasonal changes in %BF of mid-life women.

   Participant's percentage of body fat will fluctuate, and will be highest at the end of the winter season and lowest at the end of the summer season.
2. To describe predictors of seasonal changes in %BF.

There will be no intervention other than frequent monitoring of food consumption, individual activity and individual- level factors thought to influence food consumption and activity such as dietary restraint, subjective stress, sleep quality and duration, and physiological stress as measured by allostatic load. The volunteers will be asked to complete a 7-day activity and energy expenditure monitoring period (along with body composition assessment, questionnaires regarding individual factors thought to affect food consumption and activity, blood draw and urine collection to measure allostatic load) in each of the four seasons over a 12-month period; between monitoring periods they will come to the GFHNRC for measurement of weight, skin carotenoids for assessment of fruit and vegetable intake, and to provide a morning urine sample monthly (8 times), and receive emails reminding them to log on to a secure server and complete a 24-hr recall 3 times a month (36 times during the year).

The ASA-24 will be administered to assess nutritional intake; Actigraph GT3X+, Actitrainer, and QStarz GPS logger will be used to assess physical activity. Physiological stress will be assessed using the allostatic load index.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women aged 40-60 years
* Weight stable (±10 lbs) for at least 6 months prior to the start of the study
* Body mass index (BMI) between 18-35 kg/m2
* Access to high-speed internet
* Willing to comply with study requirements

Exclusion Criteria:

* BMI >35 or < 18
* Current smoker or tobacco or nicotine use
* Male sex
* Age <40.0 or >60 years
* Health conditions (cardiovascular, pulmonary, orthopedic, asthma) that would limit participation in physical activity
* Medications that would influence appetite, weight gain or weight loss.
* Intentional changes in diet or large increases in physical activity for the purpose of weight loss during the study. Typical weight maintenance behaviors are not an exclusion criterion.
* Pregnant, lactating, or planning pregnancy.
* Travel plans that do not permit full participation.
* Inability to walk without assistance. The capability to walk upright is fundamental because accelerometry measures the duration and intensity of horizontal physical activities.
* Inability to give consent.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Middle-aged females
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in body fat | Season 1, season 2, season 3, season 4
  Body fat location and amount will be assess by dual-energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA-ARS-GFHNRC
Locations (1):
- Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jahns L, Johnson LK, Conrad Z, Bukowski M, Raatz SK, Jilcott Pitts S, Wang Y, Ermakov IV, Gellermann W. Concurrent validity of skin carotenoid status as a concentration biomarker of vegetable and fruit intake compared to multiple 24-h recalls and plasma carotenoid concentrations across one year: a cohort study. Nutr J. 2019 Nov 21;18(1):78. doi: 10.1186/s12937-019-0500-0. PMID 31752882